CLINICAL TRIAL: NCT02812303
Title: Implementation of a Population Health Chronic Disease Management Program in a Primary Care Network
Brief Title: Implementation of a Population Health Chronic Disease Management Program
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Steven Atlas, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 2009P002079
Record Dates: First submitted 2016-06-20; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases; Hypertension
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Population Health Coordinator Support: 8 practices received the support of central population health coordinators (PHCs). PHCs utilized a population health management (PHM) information technology (IT) tool and performed administrative tasks including appointment scheduling, ordering overdue laboratory testing, chart reviews, and obtaining outside tests/labs. In addition, PHCs regularly met with physicians to review those patients who required clinical intervention to develop an action plan.
  The network did not have sufficient resources to implement a PHC in all of the 18 network practices. So PHCs were allocated by responses from the practice leader, baseline quality scores, size of the practice, nature of the practice (health center vs not), and location of the practice. These decisions were made in a way that sought to equitably distribute available PHC resources within the practice network as a way to get network buy-in and maximize the impact of the program, both for practices with and without PHCs.
  Interventions: Other: Centralized support for population health management activities
- No Population Health Coordinator Support: Ten practices without PHC support were provided training on how to use the PHM IT tool. The staff in these practices remained primarily responsible for managing administrative tasks.

INTERVENTIONS:
Other: Centralized support for population health management activities
  Groups: Population Health Coordinator Support

SUMMARY:
A pilot program was created by the network's primary care leadership team at Massachusetts General Hospital. A population health management program was implemented for chronic disease management. The investigators evaluated quality of care process and outcome measures over the first six months of the program and compared practices assigned a central population health coordinator to those not assigned this support.

DETAILED DESCRIPTION:
A pilot program was created by the network's primary care leadership team at Massachusetts General Hospital. They hired and allocated 4 population health coordinators (PHCs) as part of a pilot project to centralize population health management efforts to improve quality of care for chronic disease management. The network did not have sufficient resources to implement a PHC in all of the 18 network practices. So the program's team invited practice leaders to participate and the PHCs were allocated by program's leadership team based on a variety of factors including responses from the practice leader, baseline quality scores, size of the practice, nature of the practice (health center vs not), and location of the practice (on campus or community based). These decisions were made in a way that sought to equitably distribute available PHC resources within the practice network as a way to get network buy-in and maximize the impact of the program, both for practices with and without PHCs. In this study, the investigators evaluated quality of care process and outcome measures over the first six months of the chronic disease management program. The investigators hypothesized that practices assigned a central PHC would have greater performance increases in quality measures compared to practices that were not assigned a PHC.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus (type 1 or type 2), or cardiovascular disease (including coronary artery disease, peripheral vascular disease, and cerebrovascular disease), or hypertension
* Breast cancer: women 50-74 years of age
* Cervical cancer: women 21-64 years of age
* Colorectal cancer: men or women 52-75 years of age

Exclusion Criteria:

* Patients not connected with a specific network physician or practice
* Patients who switched between PHC and non-PHC practices during the follow-up period
* Breast: bilateral mastectomy
* Cervical: total hysterectomy Colorectal: total colectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult adult (age ≥ 18 years) patients who had at least one visit to a study practice within the prior 3 years at baseline or had a visit during the 6-month study evaluation period and were connected with a specific network physician or practice.
Sampling Method: Non-Probability Sample
Enrollment: 108000 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Difference in differences in Low density lipoprotein (LDL) goal achievement over the follow-up period comparing PHC to non-PHC practices | 6 months
  Among patients with diabetes and cardiovascular disease
Difference in differences in Hemoglobin A1c (HbA1c) goal achievement over the follow-up period comparing PHC and non-PHC practices | 6 months
  Among patients with diabetes
Difference in differences in Blood pressure (BP) goal achievement over the follow-up period comparing PHC and non-PHC practices | 6 months
  Among patients with diabetes and hypertension

SECONDARY OUTCOMES:
Difference in differences in proportion of patients completing breast cancer screening over the follow-up period comparing PHC and non-PHC practices | 6 months
Difference in differences in proportion of patients completing cervical cancer screening over the follow-up period comparing PHC and non-PHC practices | 6 months
Difference in differences in proportion of patients completing colorectal cancer screening over the follow-up period comparing PHC and non-PHC practices | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Atlas, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] James A, Berkowitz SA, Ashburner JM, Chang Y, Horn DM, O'Keefe SM, Atlas SJ. Impact of a Population Health Management Intervention on Disparities in Cardiovascular Disease Control. J Gen Intern Med. 2018 Apr;33(4):463-470. doi: 10.1007/s11606-017-4227-3. Epub 2018 Jan 8. PMID 29313223